CLINICAL TRIAL: NCT04690179
Title: Sarcopenia and Sarcopenic Obesity in Complex Abdominal Wall Surgery: Postoperative Complications and Their Impact on Recurrence
Brief Title: Effects of Sarcopenia and Sarcopenic Obesity in Complex Abdominal Wall Surgery
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hospital Universitario Ramon y Cajal (Other)
Responsible Party: Principal Investigator, Luis Blázquez Hernando, Surgeon, Hospital Universitario Ramon y Cajal
Other Study IDs: 1
Record Dates: First submitted 2020-12-26; First posted 2020-12-30 (Actual); Last update posted 2020-12-30 (Actual); Status verified 2020-12

CONDITIONS: Sarcopenia; Sarcopenic Obesity; Incisional Hernia
MeSH Terms: conditions — Sarcopenia; Incisional Hernia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The objective of our study is to evaluate the prevalence of sarcopenia and sarcopenic obesity in our surgical population and their relationship in postoperative complications after complex abdominal wall surgery and its influence on hernia recurrence.

This is a retrospective study on a prospective maintains database of complex abdominal wall surgery.

We select patients with defects larger than 10 cm from any location (W3 of the EHS classification), excluding other causes of complex abdominal wall in order to have a more homogeneous sample.

Pre-surgical computed tomography (CT) scans of the selected patients will be reviewed to establish the diagnosis of sarcopenia, obesity, sarcopenia-obesity or the absence of these (normal). The CT scans will be reviewed by two trained investigators, blinded to postoperative complications and survival. In case of disagreement, a third investigator will break the tie.

The radiological diagnosis of sarcopenia has been established based on the skeletal muscle mass index. Skeletal muscle mass measurement will be performed in a cross-section in the pre-surgical CT scan at the level of the third lumbar vertebra (L3).

The BMI, the Visceral Fat Area and the Subcutaneous Fat Area (SFA) will also be measured. With the previous data, the VFA / SFA ratio will be calculated.

The study will be completed with the collection of sociodemographic data, comorbidities and presence of risk factors for the development of incisional hernia, ASA, size and location of the hernia, surgical technique, postoperative complications according to Clavien-Dindo, stay, readmission, late complications and hernia recurrence. Likewise, the presence or absence of recurrence will be collected.

Statistical analysis will be performed to see if there is a correlation between sarcopenia and sarcopenic obesity with the appearance of local and systemic complications and recurrence. To evaluate the independent contribution of each variable to the presence of complications, a univariate and multivariate logistic regression analysis will be performed.

DETAILED DESCRIPTION:
The incidence of incisional hernia after laparotomy is as high as 20% according to current literature, and repair of incisional hernias is one of the most frequently performed operations by general surgeons. A not inconsiderable part of these hernias, due to their size, complexity or degree of contamination, is considered complex abdominal wall. Surgery in these patients is a major surgery that is accompanied by a marked anabolic response and a high incidence of local and systemic complications and a high recurrence rate.

In recent years, there has been a growing interest in evaluating the relationship between surgical results and body composition. Sarcopenia is a new concept that reflects the loss of skeletal muscle mass. Recent publications have recognized sarcopenia as a prognostic factor in the evolution of surgical patients operated on for cancer, transplants, trauma and emergency surgery, but there is still little evidence that it plays a role in surgery for the complex abdominal wall.

The prevalence of sarcopenia is growing progressively. One of the causes may be that life expectancy has increased worldwide and is well known that ageing is associated with the progressive loss of muscle mass (9).

Sarcopenia can be classified into primary, which is caused by ageing, and secondary, which is caused by immobility or diseases such as cancer (10).

On the other hand, obesity is defined as abnormal or excessive accumulation of fat mass. It is a major public health problem and is recognized as a risk factor for global morbidity and mortality. Its incidence continues to increase worldwide and its prevalence has doubled since 1980 (11). It is well documented that visceral obesity is associated with high complication rates in patients who undergo abdominal wall surgery (12-15).

The body mass index (BMI) has long been used to diagnose malnutrition. However, weight gain and loss are not reliable indicators of changes in body composition; generally, men store body fat in the visceral area while women store it mainly subcutaneously. Also, people tend to lose muscle mass and gain fat as they age. Therefore, patients with a similar BMI may have a different nutritional status (16).

Sarcopenic obesity combines the risks of obesity and sarcopenia and is considered the worst-case scenario (17,18).

Objectives:

The objective of our study is to evaluate the prevalence of sarcopenia and sarcopenic obesity in our population. The aim is to evaluate its relationship in postoperative complications after complex abdominal wall surgery and its influence on hernia recurrence.

Material and methods:

A retrospective study on a prospective maintains database of complex abdominal wall surgery of three hospitals.

We have decided to select only patients with defects larger than 10 cm from any location (W3 of the EHS classification) (19), excluding other causes of complex abdominal wall in order to have a more homogeneous sample (2).

Study design:

In conjunction with the Radiology Department of Ramón y Cajal University Hospital, pre-surgical computed tomography (CT) scans will be reviewed to establish the diagnosis of sarcopenia, obesity, sarcopenia-obesity or the absence of these (normal). The CT scans will be reviewed by two trained investigators, blinded to postoperative complications and survival. In case of disagreement, a third investigator will break the tie.

The radiological diagnosis of sarcopenia has been established based on the skeletal muscle mass index. Skeletal muscle mass measurement will be performed in a cross-section in the pre-surgical CT scan at the level of the third lumbar vertebra (L3). To identify muscle tissue the range -29 to +150 in Hounsfield Units (HU) will be used. The L3 region contains the following muscles: psoas, paraspinal muscles, and muscles of the abdominal wall (transverse abdominis, external and internal obliques, rectus abdominis). The skeletal muscle mass index will be calculated with the sum of the cross-sectional areas of these muscles (cm2). These values will be normalized according to the square of the patient's height (m2). As a cut-off point for the diagnosis of sarcopenia, we will use the values published by Prado et al. (≤52.4 cm2 / m2 in men and ≤38.5 cm2 / m2 for women).

To define obesity we use several indexes. The most widely accepted is body mass index (BMI)> 30 kg / m2 (25-30 kg / m2-overweight). However, this index does not take into account muscle mass and fat distribution, which are associated with different risk profiles. The Visceral Fat Area (VFA) measured by CT is strongly correlated with BMI and waist circumference. Cross-sectional measurement of VFA demonstrates a stronger correlation than anthropomorphic measurements with obesity-related conditions, such as hypertriglyceridaemia, hypertension, hyperglycemia, and low levels of high-density lipoprotein (HDL) cholesterol. The VFA measurement will be performed in a cross-section in the preoperative CT scan at the L3 level. To identify fat tissue, the range -190 to -30 in Hounsfield Units (HU) will be used.

According to the Japanese Obesity Society, we will consider visceral obesity calculated by CT as a visceral fat area (VFA)> 100cm2, regardless of sex and age. Despite the fact that the Asian population and the Western population present important differences, this data has already been used previously in European series. To complete the study, the Subcutaneous Fat Area (SFA) will also be measured. With the previous data, the VFA / SFA ratio will be calculated. The patient will be considered viscerally obese when the VFA / SFA ratio is <0.4. This correction will be used to mitigate biases derived from using values in different populations.

The study will be completed with the collection of sociodemographic data, characteristics of the surgical procedure, as well as complications derived from it. Likewise, the presence or absence of recurrence will be collected.

Study variables: sex, age, comorbidities and presence of risk factors for the development of incisional hernia, ASA, weight, height, BMI, date of surgical intervention, size and location of the hernia, surgical technique, postoperative complications according to Clavien-Dindo , stay, readmission, late complications, hernia recurrence, end-date of follow-up. To evaluate patient-reported outcomes, a quality-of-life assessment was measured preoperatively and at 1- and 2-year follow-up, using the European Registry for Abdominal Wall Hernias Quality of Life (EuraHS-QoL) score, a hernia-specific tool developed by the European Hernia Society (20). In addition, the following will be collected by radiology: skeletal muscle mass index (Skeletal Muscle Index: SMI), visceral fat area (VFA) and subcutaneous fat area (SFA).

Procedures for collecting clinical data:

First, patients potentially candidates for the study will be selected from the complex abdominal wall database of the three participating hospitals.

Data of selected patients from Hospital Ramón y Cajal will be sent to the Radiology Department of the Ramón y Cajal University Hospital for the collection of SMI, VFA and SFA in the pre-surgical CT scan.

The preoperative CT scans of the selected patients from the Henares University Hospital and the Puerta de Hierro-Majadahonda University Hospital will be recorded on a computer device to be analyzed in the Radiology Department of the Ramón y Cajal University Hospital. Once the study variables have been calculated, computing devices containing preoperative CTs will be eliminated.

Statistical analysis:

The normality of the quantitative variables will be analyzed with the Kolmogorov-Smirnov test. Continuous variables will be expressed as mean with standard deviation, and categorical variables will be represented as proportions. For comparison analysis between groups, continuous variables will be compared using the Student's t-test and categorical variables will be analyzed, as appropriate, using the χ2 test or Fisher's exact test (univariate analysis).

For the analysis of hernia recurrence, the Kaplan-Meier method will be used. In the comparison of hernia recurrence between the groups, the long-rank test will be performed. In the multivariate analysis for hernia recurrence, the Cox regression model will be used, which will include the significant variables in the univariate analysis.

To evaluate the independent contribution of each variable to the presence of complications, a univariate and multivariate logistic regression analysis will be performed with the inclusion of candidate predictors, which are significant with p <0.200 in the univariate comparison analysis.

A statistically significant result will be considered when a value of p <0.05. SPSS Statistics Version 23 will be used for statistical analysis.

Study limitations:

Retrospective study.

Schedule of activities The approval of the Clinical Research Ethics Committee of the Ramón y Cajal University Hospital is expected to be obtained in January 2021.

After this, the patients candidates to participate in the study will be selected from the complex abdominal wall data base of the three participating hospitals. We estimate that this selection will be made in the month of February.

Once the patients have been selected, the parameters described in the materials and methods section will be determined in the preoperative CT scan of each patient. We estimate that the time required to complete this part of the study will be six to eight months.

Next, a statistical analysis will be made of the data obtained from the preoperative CT scan and from the complex abdominal wall surgery database and the results will be interpreted. A manuscript will be prepared to communicate the results obtained. We estimate that this process will be performed in two or three months.

Study benefits

* To know the incidence of sarcopenia and sarcopenic obesity in complex abdominal wall patients.
* To confirm whether sarcopenia and sarcopenic obesity are risk factors for the appearance of complications and recurrence after complex abdominal wall surgery.
* This could help to better estimate the surgical risk of patients undergoing complex abdominal wall surgery.
* Sarcopenia and sarcopenic obesity are potentially modifiable with a proper nutritional and physical exercise program. If we show that sarcopenia and sarcopenic obesity are risk factors for the appearance of complications, it could help to reduce the morbidity of these patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients operated for an incisional hernia with a transverse diameter greater than 10 cm measured in the preoperative Computed Tomography.

Exclusion Criteria:

* Not having a preoperative Computed Tomography performed in the three months before the operation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing complex abdominal wall surgery at the Ramón y Cajal University Hospital, at the Puerta de Hierro-Majadahona University Hospital and at the Henares University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2021-01-18 (Estimated); Primary Completion 2021-08-15 (Estimated); Study Completion 2021-10-15 (Estimated)

PRIMARY OUTCOMES:
Complications | Thirty postoperative day
  Presence of local or systemic complications
Recurrence | Twenty four postoperative month
  Appearance of an incisional hernia recurrence

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Romain B, Renard Y, Binquet C, Poghosyan T, Moszkowicz D, Gillion JF, Ortega-Deballon P; Participating surgeons' list. Recurrence after elective incisional hernia repair is more frequent than you think: An international prospective cohort from the French Society of Surgery. Surgery. 2020 Jul;168(1):125-134. doi: 10.1016/j.surg.2020.02.016. Epub 2020 Apr 15. PMID 32305229
- [Background] Slater NJ, Montgomery A, Berrevoet F, Carbonell AM, Chang A, Franklin M, Kercher KW, Lammers BJ, Parra-Davilla E, Roll S, Towfigh S, van Geffen E, Conze J, van Goor H. Criteria for definition of a complex abdominal wall hernia. Hernia. 2014 Feb;18(1):7-17. doi: 10.1007/s10029-013-1168-6. Epub 2013 Oct 23. PMID 24150721
- [Background] Garcia-Urena MA, Lopez-Monclus J, Cuccurullo D, Blazquez Hernando LA, Garcia-Pastor P, Reggio S, Jimenez Cubedo E, San Miguel Mendez C, Cruz Cidoncha A, Robin Valle de Lersundi A. Abdominal Wall Reconstruction Utilizing the Combination of Absorbable and Permanent Mesh in a Retromuscular Position: A Multicenter Prospective Study. World J Surg. 2019 Jan;43(1):149-158. doi: 10.1007/s00268-018-4765-9. PMID 30132226
- [Background] Fukuda Y, Yamamoto K, Hirao M, Nishikawa K, Nagatsuma Y, Nakayama T, Tanikawa S, Maeda S, Uemura M, Miyake M, Hama N, Miyamoto A, Ikeda M, Nakamori S, Sekimoto M, Fujitani K, Tsujinaka T. Sarcopenia is associated with severe postoperative complications in elderly gastric cancer patients undergoing gastrectomy. Gastric Cancer. 2016 Jul;19(3):986-93. doi: 10.1007/s10120-015-0546-4. Epub 2015 Sep 25. PMID 26407875
- [Background] Peng P, Hyder O, Firoozmand A, Kneuertz P, Schulick RD, Huang D, Makary M, Hirose K, Edil B, Choti MA, Herman J, Cameron JL, Wolfgang CL, Pawlik TM. Impact of sarcopenia on outcomes following resection of pancreatic adenocarcinoma. J Gastrointest Surg. 2012 Aug;16(8):1478-86. doi: 10.1007/s11605-012-1923-5. Epub 2012 Jun 13. PMID 22692586
- [Background] Englesbe MJ, Lee JS, He K, Fan L, Schaubel DE, Sheetz KH, Harbaugh CM, Holcombe SA, Campbell DA Jr, Sonnenday CJ, Wang SC. Analytic morphomics, core muscle size, and surgical outcomes. Ann Surg. 2012 Aug;256(2):255-61. doi: 10.1097/SLA.0b013e31826028b1. PMID 22791101
- [Background] Lee JS, He K, Harbaugh CM, Schaubel DE, Sonnenday CJ, Wang SC, Englesbe MJ, Eliason JL; Michigan Analytic Morphomics Group (MAMG). Frailty, core muscle size, and mortality in patients undergoing open abdominal aortic aneurysm repair. J Vasc Surg. 2011 Apr;53(4):912-7. doi: 10.1016/j.jvs.2010.10.111. Epub 2011 Jan 7. PMID 21215580
- [Background] Englesbe MJ, Patel SP, He K, Lynch RJ, Schaubel DE, Harbaugh C, Holcombe SA, Wang SC, Segev DL, Sonnenday CJ. Sarcopenia and mortality after liver transplantation. J Am Coll Surg. 2010 Aug;211(2):271-8. doi: 10.1016/j.jamcollsurg.2010.03.039. Epub 2010 Jun 26. PMID 20670867
- [Background] Christensen K, Doblhammer G, Rau R, Vaupel JW. Ageing populations: the challenges ahead. Lancet. 2009 Oct 3;374(9696):1196-208. doi: 10.1016/S0140-6736(09)61460-4. PMID 19801098
- [Background] Santilli V, Bernetti A, Mangone M, Paoloni M. Clinical definition of sarcopenia. Clin Cases Miner Bone Metab. 2014 Sep;11(3):177-80. PMID 25568649
- [Background] Wannamethee SG, Atkins JL. Muscle loss and obesity: the health implications of sarcopenia and sarcopenic obesity. Proc Nutr Soc. 2015 Nov;74(4):405-12. doi: 10.1017/S002966511500169X. Epub 2015 Apr 27. PMID 25913270
- [Background] Nakayama M, Yoshimatsu K, Yokomizo H, Yano Y, Okayama S, Satake M, Matsumoto A, Fujimoto T, Usui T, Yamaguchi K, Shiozawa S, Shimakawa T, Katsube T, Naritaka Y. Incidence and risk factors for incisional hernia after open surgery for colorectal cancer. Hepatogastroenterology. 2014 Jul-Aug;61(133):1220-3. PMID 25436286
- [Background] Krpata DM, Blatnik JA, Novitsky YW, Rosen MJ. Evaluation of high-risk, comorbid patients undergoing open ventral hernia repair with synthetic mesh. Surgery. 2013 Jan;153(1):120-5. doi: 10.1016/j.surg.2012.06.003. Epub 2012 Aug 3. PMID 22862901
- [Background] Itatsu K, Yokoyama Y, Sugawara G, Kubota H, Tojima Y, Kurumiya Y, Kono H, Yamamoto H, Ando M, Nagino M. Incidence of and risk factors for incisional hernia after abdominal surgery. Br J Surg. 2014 Oct;101(11):1439-47. doi: 10.1002/bjs.9600. Epub 2014 Aug 14. PMID 25123379
- [Background] Aquina CT, Rickles AS, Probst CP, Kelly KN, Deeb AP, Monson JR, Fleming FJ; Muscle and Adiposity Research Consortium (MARC). Visceral obesity, not elevated BMI, is strongly associated with incisional hernia after colorectal surgery. Dis Colon Rectum. 2015 Feb;58(2):220-7. doi: 10.1097/DCR.0000000000000261. PMID 25585081
- [Background] Nishigori T, Obama K, Sakai Y. Assessment of body composition and impact of sarcopenia and sarcopenic obesity in patients with gastric cancer. Transl Gastroenterol Hepatol. 2020 Apr 5;5:22. doi: 10.21037/tgh.2019.10.13. eCollection 2020. PMID 32258526
- [Background] Prado CM, Lieffers JR, McCargar LJ, Reiman T, Sawyer MB, Martin L, Baracos VE. Prevalence and clinical implications of sarcopenic obesity in patients with solid tumours of the respiratory and gastrointestinal tracts: a population-based study. Lancet Oncol. 2008 Jul;9(7):629-35. doi: 10.1016/S1470-2045(08)70153-0. Epub 2008 Jun 6. PMID 18539529
- [Background] Muysoms FE, Miserez M, Berrevoet F, Campanelli G, Champault GG, Chelala E, Dietz UA, Eker HH, El Nakadi I, Hauters P, Hidalgo Pascual M, Hoeferlin A, Klinge U, Montgomery A, Simmermacher RK, Simons MP, Smietanski M, Sommeling C, Tollens T, Vierendeels T, Kingsnorth A. Classification of primary and incisional abdominal wall hernias. Hernia. 2009 Aug;13(4):407-14. doi: 10.1007/s10029-009-0518-x. Epub 2009 Jun 3. PMID 19495920
- [Background] Muysoms F, Campanelli G, Champault GG, DeBeaux AC, Dietz UA, Jeekel J, Klinge U, Kockerling F, Mandala V, Montgomery A, Morales Conde S, Puppe F, Simmermacher RK, Smietanski M, Miserez M. EuraHS: the development of an international online platform for registration and outcome measurement of ventral abdominal wall hernia repair. Hernia. 2012 Jun;16(3):239-50. doi: 10.1007/s10029-012-0912-7. Epub 2012 Apr 18. PMID 22527930